CLINICAL TRIAL: NCT06685692
Title: A Phase 2 Clinical Trial Investigating the Safety and Efficacy of ADX-629 in Subjects With Moderate Alcohol Associated Hepatitis
Brief Title: A Clinical Trial Investigating the Safety and Efficacy of Subjects With Alcohol Associated Hepatitis (Part 1)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADX-629-ALH-001
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Hepatitis
Keywords: ADX-629
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — ADX-629

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ADX-629 (125 mg twice daily) (Experimental)
  Interventions: Drug: ADX-629
- ADX-629 (250 mg twice daily) (Experimental)
  Interventions: Drug: ADX-629

INTERVENTIONS:
Drug: ADX-629 — 125 mg twice daily for 28 days
  Arms: ADX-629 (125 mg twice daily)
Drug: ADX-629 — 250 mg twice daily for 28 days
  Arms: ADX-629 (250 mg twice daily)

SUMMARY:
A Phase 2 Clinical Trial Investigating the Safety and Efficacy of ADX-629 in Subjects with Moderate Alcohol Associated Hepatitis (Part 1)

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 21 years old on the day of signing the informed consent form;
* Clinical diagnosis of alcoholic hepatitis, based on clinical features and laboratory testing, confirmed by the Investigator at screening
* Agreement to abstain from alcohol and utilize resources to cease at-risk behaviors during the trial, including addiction/alcohol abuse treatment
* Ability and willingness to swallow tablets
* Willingness to provide signed informed consent, prior to any trial-related procedures and willingness to comply with the trial procedures and requirements

Exclusion Criteria:

* Pregnant, intending to become pregnant (or father a child), or breastfeeding
* Current or recent enrollment in another interventional trial in the 30 days prior to screening

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Event Query | Day 1 to Day 28
  Incidence and severity of treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Synergry Healthcare, Bradenton, Florida
  - Florida Health Sciences Center/Tampa General Hospital/USF, Tampa, Florida
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - UDL Clinical Research, LLC, Houston, Texas
  - Methodist Specialty and Transplant Hospital, San Antonio, Texas
  - Bon Secours Liver Institute of Newport News, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No